CLINICAL TRIAL: NCT05720910
Title: Streamlined Geriatric and Oncological Evaluation Based on ic Technology for Holistic Patient-oriented Healthcare Management for Older Multimorbid Patients
Brief Title: Streamlined Geriatric and Oncological Evaluation Based On IC Technology
Acronym: FRONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: EUCLID Clinical Trial Platform (Other); University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IB2022-03
Record Dates: First submitted 2023-01-20; First posted 2023-02-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Comorbidities and Coexisting Conditions; Lung Cancer; Colorectal Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GERONTE (Experimental): The clinical model behind GERONTE is to regroup all health professionals taking care of a multimorbid patient, into a common care coordination pathway;
  Interventions: Other: GERONTE
- CONTROL ARM (No Intervention): Patients included in the control arm will be managed according to the standard of care.

INTERVENTIONS:
Other: GERONTE — The clinical model behind GERONTE is to regroup all health professionals taking care of a multimorbid patient, into a common care coordination pathway
  Arms: GERONTE

SUMMARY:
The primary objective of GERONTE STUDY is to evaluate the effectiveness of the GERONTE, ICT-based, integrated care pathway to improve patient 6-month quality of life, in France.

Study design is a stepped wedge randomised controlled trial. Clusters will be participating hospitals, comprising eight investigating sites in total (Figure 2).

This is a stepped wedge of cross-over type. Patients included at each "step" are different individuals. The first "step" is a reference measurement where none of the clusters will implement the intervention. The investigating sites will be randomly drawn to determine the order in which they will implement the intervention, by "steps" of two months.

The primary endpoint is the Quality of Life assessed by the EORTC QLQ-C30 (version 3.0) questionnaire at 6 months after GERONTE implementation. It has 3 sub-scores that will be analysed independently, with alpha risk adjustment.

DETAILED DESCRIPTION:
This is a stepped wedge of cross-over type. Patients included at each "step" are different individuals. The first "step" is a reference measurement where none of the clusters will implement the intervention. The investigating sites will be randomly drawn to determine the order in which they will implement the intervention, by "steps" of two months. A total of 10 patients by step are to be included in each center; these 10 patients must be regularly included along the 2-month period of each step. If 10 patients are already included before the end of the 2 months' step period, the center has to stop the inclusions till the beginning of the subsequent step. If a center, near to the end of a step, is far from reaching of the 10 patients' inclusion, it must increase the speed of its inclusions to be as close as possible of 10 patients included at the end of the step. In each center, patient sample has to be representative of type of cancer managed in the center, along the trial duration. The repartition of cancer types must be homogeneous along the steps and during the trial duration.

All participating investigating sites will have study collaborators in charge of organizing intervention implementation and data collection. The intervention will be prepared prior to the start of the trial, so that each investigating site can implement it as defined by the randomisation. Each center engaged to participate needs to participate till the end of the trial. A center commitment to participate will be requested before each center involvement to avoid center withdrawal after the start of the trial. Quantitative data regarding the myPatientSpace adapted for GERONTE app usage will be collected at each step and in each cluster by study collaborators, from the beginning of GERONTE system implementation. Care outcome data (Quality of life, anxiety, autonomy, additional hospitalisation, mortality...) will be collected by local referents at 3, 6, 9 and 12 months after inclusion in GERONTE. The data necessary to calculate the real cost of the intervention, of its implementation and of resource use data of patient management will be continuously collected during follow-up. GERONTE patient-centered system implementation and usage will be collected by the local referents in each center. Qualitative analysis will be performed in each center at GERONTE system implementation and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

- General inclusion criteria

1. Age ≥ 70 years old.
2. New or progressive cancer (breast, lung, colorectal, prostate), histologically proven or strong clinical suspicion, fulfilling the tumor specific criteria.
3. Estimated life expectancy greater than 6 months.
4. At least one moderate/severe multimorbidity inclusion criteria other than current cancer (see separate list under 5.3).
5. Patients must be willing and able to comply with study procedures.
6. Voluntarily signed and dated written informed consents prior to any study specific procedure.
7. QLQ-C30 Quality of Life Questionnaire fully completed at baseline, before inclusion.
8. Patients affiliated with a French social security scheme in accordance with the French law on biomedical research (Article 1121-11 of the French Code of Public health).

   Tumor specific inclusion criteria
9. Specific inclusion criteria for breast cancer:

   9.1. Non-metastatic breast cancer (M0):

   - No prior treatment for the current breast cancer.

   - All 3 criteria required:

   o Clinical staging: cT2-3-4 Nany, or cTany N1-2-3;
   * The cancer specialist considers* surgery;
   * The cancer specialist considers* radiotherapy and/or chemotherapy. 9.2. Metastatic breast cancer (M1): Both criteria required:

     * The cancer specialist considers* chemotherapy or PARP-inhibitors or mTOR-inhibitors / PIK3CA inhibitors; Previous endocrine therapy +/- CDK4/6 inhibitors is allowed;
     * The patient received maximum 1 prior line of chemotherapy for metastatic disease.

       * 'consider' implies that this treatment may be a treatment option for this patient in this particular setting. If at a later point, a different treatment choice is made, the patient remains eligible.
10. Specific inclusion criteria for colorectal cancer:

    10.1. Non-metastatic colorectal cancer (M0):

    - No prior therapy for the current tumor in the recruiting hospital
    * At least one of the 3 criteria required:

      o The cancer specialist considers* surgery;
      * The cancer specialist considers* radiotherapy;
      * The cancer specialist considers* chemotherapy and/or immunotherapy. 10.2. Metastatic colorectal cancer (M1):
    * The cancer specialist considers* first or second line systemic therapy and/or radiotherapy (+/- surgery). No previous chemotherapy allowed except adjuvant/perioperative chemotherapy stopped for more than 12 months.

      * 'consider' implies that this treatment may be a treatment option for this patient in this particular setting. If at a later point, a different treatment choice is made, the patient remains eligible.
11. Specific inclusion criteria for lung cancer:

11.1. Non-metastatic lung cancer (M0):

* No prior therapy for the current tumor in the recruiting hospital
* At least one of the 3 criteria required:

  * The cancer specialist considers* surgery (patients considered for treatment with percutaneous thermoablation alone are not eligible);
  * The cancer specialist considers* radiotherapy (except SBRT);
  * The cancer specialist considers* systemic therapy. Possible systemic therapies are chemotherapy and/or immune therapy and/or targeted therapy. Patients only considered* for monotherapy with anti-EGFR TKI or somatostatin analog are not eligible.

11.2. Metastatic lung cancer (M1):

* The cancer specialist considers* first or second line systemic therapy. Possible systemic therapies are chemotherapy and/or immune therapy and/or targeted therapy. Patients only considered* for monotherapy with anti-EGFR TKI or somatostatin analog are not eligible.

  *'consider' implies that this treatment may be a treatment option for this patient in this particular setting. If at a later point, a different treatment choice is made, the patient remains eligible.

  12. Specific inclusion criteria for prostate cancer: 12.1. Non-metastatic prostate cancer (M0): one of the following:
* First diagnosis M0 prostate cancer (no therapy received yet for prostate cancer): at least one of the 2 criteria required:

  o The cancer specialist considers* radiotherapy;

  o The cancer specialist considers* hormone therapy (ADT +/- combination Abiraterone and Prednisone).
* Salvage treatment M0 prostate cancer (received prior surgery at least 6 months before):

  o The cancer specialist considers* radiotherapy (+/- ADT)
* Non-metastatic castration resistant prostate cancer:

  * The cancer specialist considers* treatment intensification (ADT + Enzalutamide or Apalutamide or Darolutamide).

12.2. Metastatic prostate cancer (M1): - The cancer specialist considers* treatment with Abiraterone or Enzalutamide or Apalutamide, or Docetaxel or Cabazitaxel or PARP-inhibitors or Lutetium PSMA.

*'consider' implies that this treatment may be a treatment option for this patient in this particular setting. If at a later point, a different treatment choice is made, the patient remains eligible.

Exclusion Criteria:

1. Mental illness/cognitive impairment that limits ability to provide consent or complete trial procedures.
2. Participating to an interventional clinical trial with a non-registered anticancer drug or to another geriatric intervention trial.
3. Patients and caregivers are unable or unwilling to use ICT-devices (tablet,computer, smartphone) or the Internet according to protocol.
4. Patient already included in this study.

Ages: 70 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessed by the EORTC quality of life questionnaire (EORTC QLQ-C30 ) | 6 months
  Quality of life assessed by the quality of life questionnaire (EORTC QLQ-C30) questionnaire at 6 months after inclusion:
  * Normalised global health status score
  * Normalised score of the physical functioning scale
  * Normalised score of the emotional functioning scale the minimum value of the EORTC QLQ-C30 is 30 and the maximum value is 126, and higher scores mean a worse result.

SECONDARY OUTCOMES:
Quality of life of elders cancer patients | baseline 3, 9 and 12 months
  Scores of the quality of life questionnaire for elderly cancer patients.(QLQ-ELD14). The minimum value is 14 and the maximum value is 40, and higher scores mean a worse result.
Quality of life by the EORTC quality of life questionnaire (EORTC QLQ-C30 ) | baseline 3, 9 and 12 months
  The quality of life questionnaire (QLQ-C30) scores. The minimum value of the EORTC QLQ-C30 is 30 and the maximum value is 126, and higher scores mean a worse result.
Survival | at 12 months
  Overall survival and progression-free survival
Patient frailty | baseline, 3, 6, 9 and 12 months
  Score of the Clinical frailty scale
Patient autonomy, | baseline, 3, 6, 9 and 12 months
  Dependence score of the Activities of Daily Living scale (ADL); Proportion of patients living at home; Number of completed chair stands in 30 seconds
Patient weight evolution | baseline, 3, 6, 9 and 12 months
  Weight in Kilograms
Patient anxiety | baseline, 3, 6, 9 and 12 months
  Score of Hospital Anxiety and Depression (HAD) scale. The minimum value is 0 and the maximum value is 21, and higher scores mean a worse result.
institutionalisation | 6 and 12 months
  Proportion of patient institutionalised per participants
unscheduled hospitalisations | 6 and 12 months
  Proportion of unscheduled hospitalisations per participants
Cost per life years gained | baseline, 3, 6, 9 and 12 months
  using utility assessed through normalised scores of EQ-5D-5L questionnaire
Caregiver burden in health, psychological well-being, finances, social life and relationship with patient | baseline, 3, 6, 9 and 12 months
  Zarit Burden Interview
Patient experience of person-centered coordinated care | 6 and 12 months
  Person-Centered Coordinated Care Experience Questionnaire (P3CEQ)The minimum value is 0 and the maximum value is 45, and higher scores mean a better result.
Patient, physician and health-professionals-reported overall satisfaction with the IC technology of the GERONTE system | 6 and 12 months
  Score derived from the mHealth App Usability Questionnaire (MAUQ) for standalone mHealth Apps using the Patient version for patient satisfaction and the provider version for physician and health-professional.The minimum value is 0 and the maximum value is 126, and higher scores mean a better result.
GERONTE patient-centered system implementation and usage | 6 months
  use of the myPatientSpace adapted for GERONTE app measures, for instance: number and frequency of connections.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Léon Bérard, Lyon
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Hospitalier Universitaire de Nice, Nice
  - Centre Antoine Lacassagne, Nice
  - Hôpital Tenon AP-HP, Paris
  - Centre Eugène Marquis, Rennes
  - Groupe Hospitalier Rance Emeraude, St-Malo

REFERENCES:
- [Derived] Hamaker ME, Wildiers H, Ardito V, Arsandaux J, Barthod-Malat A, Davies P, Degol L, Ferrara L, Fourrier C, Kenis C, Kret M, Lalet C, Pelissier SM, O'Hanlon S, Rostoft S, Seghers N, Saillour-Glenisson F, Staines A, Schwimmer C, Thevenet V, Wallet C, Soubeyran P. Study protocol for two stepped-wedge interventional trials evaluating the effects of holistic information technology-based patient-oriented management in older multimorbid patients with cancer: The GERONTE trials. J Geriatr Oncol. 2024 May;15(4):101761. doi: 10.1016/j.jgo.2024.101761. Epub 2024 Apr 5. PMID 38581958